CLINICAL TRIAL: NCT01248910
Title: SASES: SAlzburg Skiing in the Elderly Study: Health Benefits of Alpine Skiing for the Elderly
Brief Title: Health Benefits of Alpine Skiing for the Elderly
Acronym: SASES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salzburg (Other)
Collaborators: Manchester Metropolitan University (Other); University of Freiburg (Other); University of Copenhagen (Other); Paracelsus Medical University (Other)
Responsible Party: Erich Müller, Department of Sport Science and Kinesiology, University of Salzburg
Other Study IDs: SASES
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-10

CONDITIONS: Elderly; Strength; Exercise Capacity; Postural Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpine Skiing (Experimental)
  Interventions: Behavioral: Alpine Skiing
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Alpine Skiing
  Arms: Alpine Skiing

SUMMARY:
Older people tend to live a sedentary lifestyle which causes a loss of cardiorespiratory fitness, impaired postural stability and a increased risk of falls. Social isolation of older people leads to depression and other mental diseases. However, numerous studies show that age-related degradation processes and functional limitations can be counteracted by physical activity. Various studies show that alpine skiing is a complex sport that places demands on the cardiorespiratory, neuromuscular and sensorimotor systems. With studies providing evidence to suggest alpine skiing is an appropriate activity for elderly as a health-enhancing sport, perhaps Alpine skiing could provide the physical activity needed to counteract age-related degradation processes and loss of function. To date, there is a lack of long-term intervention studies devoted to this topic. The aim of this study was to monitor the long-term effects of skiing on the health of older people, as to age-related muscle breakdown, cardiorespiratory fitness, body stability, general mobility and the overall psychological state of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-75 years of age at
* average or above average skiing ability
* average physical activity level
* willingness to ski regularly (2-3 days per week) for 12 weeks
* ability to give written informed consent

Exclusion Criteria:

* serious health problems that would make alpine skiing unjustifiable

Ages: 60 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erich Müller, PhD, Principal Investigator — Department of Sport Science and Kinesiology, University of Salzburg
Locations (1):
- Department of Sport Science and Christian Doppler Laboratory "Biomechanics in Skiing", Hallein, Salzburg, Austria